CLINICAL TRIAL: NCT03647696
Title: Incidence of Opioid-induced Respiratory Depression in Medical and Trauma Patients on the General Care Floor Receiving Patient-controlled Analgesia and Nurse Administered Intravenous Opioids Monitored by Capnography and Pulse Oximetry: A Prospective, Blinded Observational Study
Brief Title: Incidence of Opioid-Induced Respiratory Depression in Medical and Trauma Patients
Status: Withdrawn | Type: Observational
Why Stopped: Principal Investigator left institution and took the study them.
Sponsor: Poudre Valley Health System (Other)
Collaborators: University of Colorado Health (Other); University of California, Los Angeles (Other); Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: PoudreVHS
Record Dates: First submitted 2018-08-22; First posted 2018-08-27 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Respiratory Depression; Sedation
Keywords: respiratory depression, opioid-induced sedation
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of this prospective, blinded observational study is to correlate assessment of sedation and respiratory status with capnography and pulse oximetry monitoring in hospitalized adult medical and trauma patients receiving patient-controlled analgesia (PCA) or nurse administered intravenous (IV) opioids for acute pain. Nursing assessment of respiratory status and sedation level will be correlated with capnography and pulse oximetry values as technology-supported monitoring to identify respiratory depression and opioid-induced sedation. The secondary objective is to identify capnography and pulse oximetry values that correlate with respiratory decompensation and opioid-induced sedation in medical and trauma patients on the general care floor.

ELIGIBILITY:
Inclusion Criteria:

1. Spontaneously breathing adults 18 to 89 years of age
2. English speaking
3. Receiving PCA or nurse administered IV opioids for medical or trauma-related pain
4. Admitted to the general care floor from the emergency department

Exclusion Criteria:

1. Less than 18 or greater than 89 years of age
2. Transfer to the general care floor from the Intensive Care Unit
3. Receiving intrathecal or epidural opioids
4. Inability or unwillingness to wear the etCO2 sampling line nasal cannula or pulse oximetry sensor
5. History or diagnosis of a sleep disordered breathing syndrome
6. Use of Continuous Positive Airway Pressure or (CPAP) or Bilevel Positive Airway Pressure (BIPAP) non-invasive ventilation as home regime
7. Receiving non-invasive ventilation
8. Presence of a co-morbidity that impacts respiration or ventilation (e.g Chronic Obstructive Pulmonary Disease or Pulmonary Fibrosis)
9. Unwilling or unable to participate
10. Member of a vulnerable population such as pregnant women or prisoners.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target study population will be hospitalized, adult medical or trauma patients on the general care floor receiving PCA or nurse administered IV opioids for acute pain.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Hypoventilation | Change from baseline measurement observed within 60 minutes after opioid administration
  Continuous respiratory monitoring using capnography will be performed for collecting data of end-tidal carbon dioxide (etCO2)

SECONDARY OUTCOMES:
Hypoxemia | Change from baseline measurement observed within 60 minutes after opioid administration
  Continuous respiratory monitoring using pulse oximetry will be performed for collecting data of oxygen saturation (SpO2)

OTHER OUTCOMES:
Sedation | Change from baseline assessment observed within 60 minutes after opioid administration
  Sedation assessment will be preformed using the Moline-Roberts Pharmacologic Sedation Scale in which sedation levels of 1, 2, 3, 4, 5, 6 are assessed where increasing numbers represent increasing levels of Sedation and sedation levels 3 or 4 or 5 or 6 indicate unintended opioid-induced sedation for the purpose of this study
Sedation | Change from baseline assessment observed with 60 minutes after opioid administration
  Sedation assessment will be preformed using the Pasero Opioid-Induced Sedation Scale in which sedation levels of S, 1, 2, 3, 4 are assessed where "S" represents normal sleep and increasing numbers represent increasing levels of Sedation and sedation levels 3 or 4 indicate unintended opioid-induced sedation for the purpose of this study

CONTACTS AND LOCATIONS:
Overall Officials: Susan J Dempsey, PhD(c), Principal Investigator — UCLA and UCHealth

IPD SHARING:
Plan to Share IPD: Undecided
It is not decided whether the data will be available for sharing

REFERENCES:
- [Background] Sun Z, Sessler DI, Dalton JE, Devereaux PJ, Shahinyan A, Naylor AJ, Hutcherson MT, Finnegan PS, Tandon V, Darvish-Kazem S, Chugh S, Alzayer H, Kurz A. Postoperative Hypoxemia Is Common and Persistent: A Prospective Blinded Observational Study. Anesth Analg. 2015 Sep;121(3):709-715. doi: 10.1213/ANE.0000000000000836. PMID 26287299
- [Background] Stites M, Surprise J, McNiel J, Northrop D, De Ruyter M. Continuous Capnography Reduces the Incidence of Opioid-Induced Respiratory Rescue by Hospital Rapid Resuscitation Team. J Patient Saf. 2021 Sep 1;17(6):e557-e561. doi: 10.1097/PTS.0000000000000408. PMID 28731933
- [Background] Perman SM, Stanton E, Soar J, Berg RA, Donnino MW, Mikkelsen ME, Edelson DP, Churpek MM, Yang L, Merchant RM; American Heart Association's Get With the Guidelines(R)-Resuscitation (formerly the National Registry of Cardiopulmonary Resuscitation) Investigators. Location of In-Hospital Cardiac Arrest in the United States-Variability in Event Rate and Outcomes. J Am Heart Assoc. 2016 Sep 29;5(10):e003638. doi: 10.1161/JAHA.116.003638. PMID 27688235
- [Background] Churpek MM, Yuen TC, Huber MT, Park SY, Hall JB, Edelson DP. Predicting cardiac arrest on the wards: a nested case-control study. Chest. 2012 May;141(5):1170-1176. doi: 10.1378/chest.11-1301. Epub 2011 Nov 3. PMID 22052772
- [Background] Andersen LW, Berg KM, Chase M, Cocchi MN, Massaro J, Donnino MW; American Heart Association's Get With The Guidelines((R))-Resuscitation Investigators. Acute respiratory compromise on inpatient wards in the United States: Incidence, outcomes, and factors associated with in-hospital mortality. Resuscitation. 2016 Aug;105:123-9. doi: 10.1016/j.resuscitation.2016.05.014. Epub 2016 May 30. PMID 27255952
- [Background] Lee LA, Caplan RA, Stephens LS, Posner KL, Terman GW, Voepel-Lewis T, Domino KB. Postoperative opioid-induced respiratory depression: a closed claims analysis. Anesthesiology. 2015 Mar;122(3):659-65. doi: 10.1097/ALN.0000000000000564. PMID 25536092
- [Background] Jarzyna D, Jungquist CR, Pasero C, Willens JS, Nisbet A, Oakes L, Dempsey SJ, Santangelo D, Polomano RC. American Society for Pain Management Nursing guidelines on monitoring for opioid-induced sedation and respiratory depression. Pain Manag Nurs. 2011 Sep;12(3):118-145.e10. doi: 10.1016/j.pmn.2011.06.008. PMID 21893302
- [Background] Taenzer AH, Pyke JB, McGrath SP, Blike GT. Impact of pulse oximetry surveillance on rescue events and intensive care unit transfers: a before-and-after concurrence study. Anesthesiology. 2010 Feb;112(2):282-7. doi: 10.1097/ALN.0b013e3181ca7a9b. PMID 20098128
- [Background] Taenzer AH, Pyke J, Herrick MD, Dodds TM, McGrath SP. A comparison of oxygen saturation data in inpatients with low oxygen saturation using automated continuous monitoring and intermittent manual data charting. Anesth Analg. 2014 Feb;118(2):326-331. doi: 10.1213/ANE.0000000000000049. PMID 24361847
- [Background] Davis C, Geik C, Arthur K, Fuller J, Johnston E, Levitt F, Leung E, McCart G, McMichael D, Painter J, Staublin T, Walroth T. A Multisite Retrospective Study Evaluating the Implementation of the Pasero Opioid-Induced Sedation Scale (POSS) and Its Effect on Patient Safety Outcomes. Pain Manag Nurs. 2017 Aug;18(4):193-201. doi: 10.1016/j.pmn.2017.03.006. Epub 2017 Jun 9. PMID 28606595
- [Background] Morris TA, Gay PC, MacIntyre NR, Hess DR, Hanneman SK, Lamberti JP, Doherty DE, Chang L, Seckel MA. Respiratory Compromise as a New Paradigm for the Care of Vulnerable Hospitalized Patients. Respir Care. 2017 Apr;62(4):497-512. doi: 10.4187/respcare.05021. PMID 28341777
- [Background] Henneman EA, Gawlinski A, Giuliano KK. Surveillance: A strategy for improving patient safety in acute and critical care units. Crit Care Nurse. 2012 Apr;32(2):e9-18. doi: 10.4037/ccn2012166. PMID 22467622
- [Background] Moline B, Roberts M, Houser J. Validity and interrater reliability of the Moline-Roberts Pharmacologic Sedation Scale. Clin Nurse Spec. 2012 May-Jun;26(3):140-8. doi: 10.1097/NUR.0b013e3182503fd6. PMID 22504472
- [Background] Overdyk FJ, Carter R, Maddox RR, Callura J, Herrin AE, Henriquez C. Continuous oximetry/capnometry monitoring reveals frequent desaturation and bradypnea during patient-controlled analgesia. Anesth Analg. 2007 Aug;105(2):412-8. doi: 10.1213/01.ane.0000269489.26048.63. PMID 17646499